CLINICAL TRIAL: NCT06465082
Title: Role of Diaphragmatic Thickening Fraction as a Predictor of Successful Weaning From Mechanical Ventilation
Brief Title: Diaphragmatic Thickening Fraction as a Predictor of Successful Weaning
Status: Recruiting | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine, Mansoura University Hospital
Other Study IDs: R.24.05.2632
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: mechanical ventilation.; diaphragmatic thickening Fraction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the validity of the diaphragmatic thickening Fraction measured by ultrasound as a predictor for successful weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Timing is critical for proper weaning for patients undergoing mechanical ventilation; if this is performed prematurely complications can include increased cardiovascular and respiratory stress, CO2 retention and hypoxemia. However, unnecessary delay in weaning can also cause a number of side-effects.Weaning outcomes have been assessed by several indices. Variables such as minute ventilation, Pao2/Fio2, rapid shallow breathing index and static compliance have all been used, with variable predictive values. Previous studies have proved that diaphragmatic dysfunction is one of the main etiologies of difficult weaning, because the diaphragm progressively weakens with mechanical ventilation.Methods used to assess diaphragm function, such as fluoroscopy, phrenic nerve stimulation, measurement of trans-diaphragmatic pressure and dynamic magnetic resonance imaging of the diaphragm, all have limitations. These include ionizing radiation exposure, low availability, invasiveness and necessity for patient transportation. Conversely, the use of ultrasound is safe, non-invasive, avoids radiation side-effects, and is available at the bedside.The aim of this study is to assess the validity of the diaphragmatic thickening Fraction measured by ultrasound as a predictor for successful weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years old, who are in need for mechanical ventilation as: Life threatening hypoxia, Respiratory rate > 30 breath/min, Disturbed conscious level.

Exclusion Criteria:

* Age <18 years.
* Pregnancy
* Surgical incisions likely to interfere with ultrasound examination.
* Hepato-splenomegaly, Ascites
* Neuromuscular disease as Myasthenia gravis, kypho-scoliosis
* Diaphragmatic Paralysis (paralyzed diaphragm exhibiting abnormal paradoxical movement, i.e., moving in a cranial direction during inspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients >18 years old, who are in need for mechanical ventilation as: Life threatening hypoxia, Respiratory rate > 30 breath/min, Disturbed conscious level.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic thickening Fraction as predictor for weaning from mechanical ventilation. | Baseline and after 6 month
  assess the validity of the diaphragmatic thickening Fraction measured by ultrasound as a predictor for successful weaning from mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Mansoura University
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt